CLINICAL TRIAL: NCT01477840
Title: Phase 2-3 Study of Comparative of Effects of Sublingual Misoprostol and Infusion Oxytocin in Reduction of Blood Loss at Cesarean Deliveries
Brief Title: Comparative of Effects of Sublingual Misoprostol and Infusion Oxytocin in Reduction of Bleeding at Cesarean
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soudabeh Eshghi ali (Other)
Collaborators: Kermanshah University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Soudabeh Eshghi ali, Obstetrics & Gynecology Department, Kermanshah University of Medical Sciences
Organization: Kermanshah University of Medical Sciences (Other)
Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Kermanshah University
Record Dates: First submitted 2011-10-31; First posted 2011-11-23 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Bleeding Intraoperative
Keywords: Misoprostol; Oxytocin; Cesarean Delivery; Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Misoprostol (Experimental)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Sublingual Misoprostol 200 Micrograms After Spinal Anesthesia
  Other Names: Brand Name: Cytotec, Cyotec, Serial 022-00 , Code A02BB01

SUMMARY:
The purpose of this study is to determine whether the effect of sublingual misoprostol is better than infusion oxytocin in reduction of blood loss at cesarean deliveries.

DETAILED DESCRIPTION:
A total of 180 pregnant women with gestational age 37 weeks and over who underwent cesarean operation in Imam Reza hospital had elective or emergency procedure with incision in lower segment during one year recruitment. The patients were randomly assigned to undergo 200 micrograms misoprostol sublingual or 400 micrograms and infusion 20 unit oxytocin after spinal anesthesia. Main outcome measures: The length of surgery, bleeding volume, the need for transfusion, fever, tachycardia, and hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Indication of Cesarean Deliveries
* Elective or Emergency with Incision in Lower Segment in Women with
* Gestational Age more than 37 Weeks.

Exclusion Criteria:

* Anemia
* Multiple Pregnancy
* Polyhydraminus
* Prolonged Labor
* Premature Rupture of Membrane and Patients had Previous History of Diabetes Mellitus
* Hypertension
* Cardiovascular Disease
* Coagulopathy Disease

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Intraoperative bleeding | At the time of surgery

SECONDARY OUTCOMES:
Fever | During 48 hours after surgery measured every 3 hours
Changing of pulse rate from base | Before surgery & intraoperative & 6 hours after surgery
Changing of blood pressure | Before surgery & intraoperative & 6 hours after surgery
Diarrhea | Before & 6 hours after surgery
Vomiting | Before & 6 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anisodowleh Nankali, MD, Study Chair — Kermanshah University of Medical Sciences
Locations (1):
- KUMS Obstetrics & Gynecology Department, Imam Reza Hospital, Kermanshah, Kermanshah Province, Iran

REFERENCES:
- [Result] Eftekhari N, Doroodian M, Lashkarizadeh R. The effect of sublingual misoprostol versus intravenous oxytocin in reducing bleeding after caesarean section. J Obstet Gynaecol. 2009 Oct;29(7):633-6. doi: 10.1080/01443610903061744. PMID 19757270